CLINICAL TRIAL: NCT03803670
Title: Clinical Significance of Occult Central Nervous System Disease In Adult Acute Lymphoblastic Leukemia: A Multicenter, Retrospective Study From The Campus All/Gimema Network
Brief Title: Clinical Significance of Occult Central Nervous System Disease In Adult Acute Lymphoblastic Leukemia
Status: Completed | Type: Observational
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Maria Ilaria Del Principe, PI, University of Rome Tor Vergata
Other Study IDs: RS176/17
Record Dates: First submitted 2019-01-10; First posted 2019-01-14 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: acute lymphoblastic leukemia; flow cytometry
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- acute lymphoblastic leukemia patients: We observed within adult patients with ALL three groups of patients: patients without central nervous system (CNS) involvement, patients with manifest CNS involvement and patients with occult CNS involvement.
  Interventions: Diagnostic Test: evaluation of cerebrospinal fluid of ALL

INTERVENTIONS:
Diagnostic Test: evaluation of cerebrospinal fluid of ALL — We evaluated cerebrospinal fluids of patients with ALL by conventional cytology and by flow cytometry

SUMMARY:
Central nervous system involvement at diagnosis remains an obstacle to a long-term cure of patients affected by acute lymphoblastic leukemia. The investigators have previously reported that flow cytometry (FCM) is better than conventional cytology (CC) in demonstrating the presence of leukemic cells in the patients'(pts) cerebrospinal fluid (CSF), especially in samples with low cell counts. In the framework of the national Campus ALL program aimed at improving the management of adult ALL patients in the context of the GIMEMA protocols, in the present study the investigators retrospectively evaluated the incidence of occult CNS positivity and its impact on outcome in 241 adult pts with newly diagnosed ALL from 13 centers.

DETAILED DESCRIPTION:
Demographic and of laboratory data of 241 adult patients with ALL were retrospectively recorded. All patients underwent diagnostic lumbar puncture and each cerebrospinal fluid sample was examined by CC and FCM. The investigators identified patients with the only FCM positivity and the investigators correlated this condition with clinical and of laboratory data and with clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* ALL at onset
* Age >18 years

Exclusion Criteria:

* ALL relapsed or refractory
* Age <18 years

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients affected by ALL underwent to diagnostic lumbar puncture
Sampling Method: Non-Probability Sample
Enrollment: 241 (Actual)
Dates: Start 2007-01-01; Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
impact of occult CNS disease | 10 years
  relapse rate
impact of occult CNS disease on outcome | 10 years
  overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Maria Ilaria Del Principe, MD, Principal Investigator — University Tor Vergata of Rome

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Del Principe MI, Buzzatti E, Piciocchi A, Forghieri F, Bonifacio M, Lessi F, Imbergamo S, Orciuolo E, Rossi G, Fracchiolla N, Trappolini S, Neri B, Sarlo C, Zappasodi P, Dargenio M, Cefalo M, Irno-Consalvo MA, Conti C, Paterno G, De Angelis G, Sciume M, Della Starza I, Venditti A, Foa R, Guarini AR. Clinical significance of occult central nervous system disease in adult acute lymphoblastic leukemia. A multicenter report from the Campus ALL Network. Haematologica. 2021 Jan 1;106(1):39-45. doi: 10.3324/haematol.2019.231704. PMID 31879328